CLINICAL TRIAL: NCT02143778
Title: Clinical Study of the BreathID® LF System to Train the Algorithm for the ¹³C-Methacetin Breath Test (MBT) in Assessment of Portal Hypertension in Patients With Compensated Liver Cirrhosis
Brief Title: Assessing Portal Hypertension With Methacetin Breath Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSPH-EX-4014; 2014-002037-59 (EudraCT Number)
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Patients With Compensated Liver Cirrhosis
Keywords: MBT; CSPH; HVPG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compensated cirrhotic patients (Experimental): A methacetin breath test will be performed on patients who are undergoing the HVPG procedure due to their clinical indication of compensated cirrhosis.
  Interventions: Device: Methacetin Breath Test

INTERVENTIONS:
Device: Methacetin Breath Test — 13C labelled methacetin solution for breath test monitoring

SUMMARY:
This study will be used to train an algorithm using Methacetin breath test (MBT) measures and to select a cut-off to determine presence or absence of Clinically Significant Portal Hypertension (CSPH) as defined by Hepatic Venous Gradient Pressure (HVPG) ≥ 10mmHg,

DETAILED DESCRIPTION:
The portal pressure leaving the liver is measured by using a balloon catheter before and after a wedge. The difference of the pressure between the wedge and the free is the hepatic venous pressure gradient. Methacetin breath test is hypothesized to also identify CSPH and the agreement to the reference standard (HVPG) will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women (>18 years of age)
* Known chronic liver disease with cirrhosis
* Europe: Indicated to undergo HVPG testing
* US: Consented for HVPG
* For patients treated with beta blockers: They have to be on a stable dose for at least 6 weeks prior to any study related tasks
* For patients who stopped their treatment with beta blockers: Their last dose should be at least 6 weeks prior to any study related tasks

Exclusion Criteria:

* Decompensated cirrhosis as clinically defined by the presence of ascites, hepatic encephalopathy, variceal bleeding or hepatorenal syndrome
* Renal failure (creatinine > 2.5 mg/dl)
* Known acute renal tubular disease Known hypotension (Systolic Pressure <100mmHg)
* Hypocoagulablity defined as PT >6 and INR >2.3.
* Congestive heart failure (assessed clinically as NIHA >2)
* Known pulmonary hypertension (right ventricular systolic pressure > 45 mm Hg)
* Uncontrolled diabetes mellitus (HBA1C >9.5gr%)
* Concurrent prednisone or immunosuppressive treatment, if therapy and/or response to treatment are not stable for at least 3 months.
* Documented or suspected hepatocellular carcinoma
* Gastric bypass surgery or extensive small bowel resection
* Total parenteral nutrition
* Any organ transplant recipient
* Pregnant or breast feeding
* Allergy to acetaminophen and/or other related medications
* Documented drug-related concurrent hepatotoxicity or drug-related silent steatosis or drug-related fibrosis (e.g. amiodarone, methotrexate and tamoxifen)
* Uncontrolled malabsorption or diarrhea
* Documented non-cirrhotic PHT, partial / complete portal venous occlusion, hepatic venous occlusion, previous PHT surgery, or placement of a transjugular intrahepatic portosystemic shunt (TIPS)
* Primary or secondary biliary cirrhosis, primary or secondary sclerosing cholangitis, hepatic sarcoidosis, or other cholestatic disorders
* Subjects unable to perform the MBT within 7 days of HVPG procedure.
* Subject should not have taken any of the following for at least 48 hours prior to the breath test: Acyclovir , allopurinol, amiodarone, carbamazepine, cimetidine, ciprofloxacin, daidzein, (herbal) disulfiram, echinacea, enoxacin, famotidine, fluvoxamine, methoxsalen, mexiletine, montelukast, norfloxacin, phenylpropanolamine, phenytoin, propafenone, rifampin, terbinafine, ticlopidine, thiabendazole, verapamil, zileuton or oral contraceptives or any medication that might interfere with Methacetin metabolism or might affect CYP 1A2
* Subject should not have taken amiodarone or statins within the last 30 days prior to the breath test or HVPG procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Garcia Pagan, MD, Principal Investigator — University Hospital Barcelona
Locations (8):
- United States (3):
  - VA Connecticut HealthCare System, New Haven, Connecticut
  - Duke University Medical Center, Durham, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia
- France (2):
  - Hôpital Beaujon, Paris
  - Hopital Purpan, Toulouse
- Spain (2):
  - (University of Barcelona) Hospital Clinic, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
- Inselspital, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Compensated Cirrhotic Patients
Started | 246
Completed | 243
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Device malfunction | 1

BASELINE CHARACTERISTICS:
Arm/Group | Compensated Cirrhotic Patients
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 242
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39
  France | 40
  Switzerland | 9
  Spain | 158

OUTCOME MEASURES:

1. Primary Outcome: CSPH (Clinically Significant Portal Hypertension)
Description: Clinically significant portal hypertension is defined as Hepatic Venous Pressure Gradient (HVPG)>=10mmHg, whereby the portal pressure leaving the liver is measured by using a balloon catheter before and after a wedge. The difference of the pressure between the wedge and the free is the hepatic venous pressure gradient. Methacetin breath test is hypothesized to also identify CSPH and the agreement to the reference standard (HVPG) will be assessed in this study.
Time Frame: 1 hour
Population: Compensated cirrhotic patients with CSPH based on breath test compared to CSPH from HVPG (reference standard)
Measure: Mean (95% Confidence Interval); unit: percentage of agreement
Groups:
- Compensated Cirrhotic Patients With CSPH: A methacetin breath test will be performed on patients who are undergoing the HVPG procedure due to their clinical indication of compensated cirrhosis.
  Methacetin Breath Test: 13C labelled methacetin solution for breath test monitoring
Arm/Group | Compensated Cirrhotic Patients With CSPH
Number analyzed (Participants) | 246
percentage of agreement | 81.82 [74.22 to 89.42]

2. Secondary Outcome: Hepatic Venous Pressure Gradient (HVPG)>=12; Severe Portal Hypertension (SPH)
Description: Hepatic Venous Pressure Gradient greater than 12 (SPH) is an indicator of bleeding varices. whereby the portal pressure leaving the liver is measured by using a balloon catheter before and after a wedge. The difference of the pressure between the wedge and the free is the hepatic venous pressure gradient. Methacetin breath test is hypothesized to also identify SPH and the agreement to the reference standard (HVPG) will be assessed in this study.
Time Frame: 1 hour
Population: Compensated cirrhotic Patients with Severe Portal Hypertension based on MBT compared to HVPG (reference standard)
Measure: Mean (95% Confidence Interval); unit: percentage of agreement
Groups:
- Compensated Cirrhotic Patients With SPH: A methacetin breath test will be performed on patients who are undergoing the HVPG procedure due to their clinical indication of compensated cirrhosis with severe portal hypertension.
  Methacetin Breath Test: 13C labelled methacetin solution for breath test monitoring
Arm/Group | Compensated Cirrhotic Patients With SPH
Number analyzed (Participants) | 246
percentage of agreement | 76.39 [66.58 to 86.20]

ADVERSE EVENTS:
Time Frame: The Methacetin used in the breath test has a high extraction rate and is removed after less than 48 hours. Follow up was done for 48 hours after breath test. After 30 days another follow up phone call was made.
Arm/Group | Compensated Cirrhotic Patients
All-Cause Mortality (participants affected / at risk) | 0/246
Serious Adverse Events (participants affected / at risk) | 1/246
Other Adverse Events (participants affected / at risk) | 2/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compensated Cirrhotic Patients (N=246)
Severe Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compensated Cirrhotic Patients (N=246)
UTI (Infections and infestations) | 2 (2) — Urinary Tract Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT02143778/Prot_SAP_000.pdf